CLINICAL TRIAL: NCT06166316
Title: Effect of Implant Position on Clinical Outcomes of Implant-retained Mandibular Overdenture. A 3-year Retrospective Study
Brief Title: Effect of Implant Position on Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01011023RP
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Bone Loss; Patient Satisfaction
Keywords: peri-implant; retention; overdenture; patient satisfaction
MeSH Terms: conditions — Bone Diseases, Metabolic; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lateral incisor group (Active Comparator): patients having mandibular two implants in lateral incisor positions.
  Interventions: Device: overdenture retained by locator attachments.
- canine group (Active Comparator): patients having mandibular two implants in the canine positions.
  Interventions: Device: overdenture retained by locator attachments.
- premolar group (Active Comparator): patients having mandibular two implants in the premolar positions.
  Interventions: Device: overdenture retained by locator attachments.

INTERVENTIONS:
Device: overdenture retained by locator attachments. — • Implant-retained overdenture construction procedures:
  1. Primary maxillary and mandibular impressions were made, and custom trays were fabricated using auto-polymerizing acrylic resin.
  2. Definitive impressions were made with non-eugenol zinc oxide paste, and the impression copings were threaded to the implants, and polyether material was injected around the copings through the opening of the tray. Auto-polymerizing acrylic resin was used to pick up the copings with the tray. Implant analogs were screwed to the copings and the impressions was poured with stone.
  3. Locator abutment (Dentium, Co. Ltd., Korea) screwed in the analogs. Jaw relations were recorded, and semi-anatomical acrylic teeth eeee arranged in balanced occlusion.
  4. The locator housing and retentive clips were incorporated into the fitting surface of the overdentures during denture processing.

SUMMARY:
the study aims to investigate the clinical influence of different implant locations; lateral incisor, canine, and first premolar areas; supporting 2-implant retained mandibular over-dentures with locator attachment on prosthesis retention and peri-implant health.

DETAILED DESCRIPTION:
the study aims to investigate the clinical influence of different implant locations; lateral incisor, canine, and first premolar areas; supporting 2-implant retained mandibular over-dentures with locator attachment on prosthesis retention and peri-implant health.

* Thirty-six edentulous patients will be recalled from the database set of the clinic of the removable prosthodontic department, Faculty of Dentistry, Mansoura University. Patients will be recruited from previous studies, having two-implant mandibular overdentures.
* All selected patients with the following criteria: mandibular two implants retained overdenture opposing complete edentulous maxillary arch, attended the previous follow-up recalls with previous CBCT examination. Patients who didn't attend previous follow-up recalls, didn't perform radiographic follow-up, or had para-functional habits will be excluded from the study.
* The patients will be grouped based on the implant position:

Group I (12 patients): patients having mandibular two implants in lateral incisor positions.

Group II (12 patients): patients having mandibular two implants in the canine positions.

Group III (12 patients): patients having mandibular two implants in the premolar positions.

* Implant-retained overdenture construction procedures:

  1. Primary maxillary and mandibular impressions were made, and custom trays were fabricated using auto-polymerizing acrylic resin. The mandibular tray was fabricated with holes above the implant sites and molded with green impression compound modeling plastic.
  2. Definitive impressions were made with non-eugenol zinc oxide paste, and the impression copings were threaded to the implants, and polyether material was injected around the copings through the opening of the tray. Auto-polymerizing acrylic resin was used to pick up the copings with the tray. Implant analogs were screwed to the copings and the impressions was poured with stone.
  3. Locator abutment (Dentium, Co. Ltd., Korea) screwed in the analogs. Jaw relations were recorded, and semi-anatomical acrylic teeth eeee arranged in balanced occlusion.
  4. The locator housing and retentive clips were incorporated into the fitting surface of the overdentures during denture processing.

     Method of evaluation
* Assessment of the peri-implant soft tissue health including Plaque index, Probing depth, and bleeding index. Also, evaluation of the peri-implant bone loss was done at one, two, and three years after insertion using a CBCT, following the methodology described by Elsyad et al.
* Measurements of retention values: using the device of measuring the clinical retentive forces.
* Assessment of patient satisfaction and Oral Health-Related Quality of Life: using a visual analog scale (VAS) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* mandibular two implants retained overdenture opposing complete edentulous maxillary arch.
* patients who attended the previous follow-up recalls with previous CBCT examination

Exclusion Criteria:

* Patients who didn't attend previous follow-up recalls.
* patients who didn't perform radiographic follow-up.
* patients who had para-functional habits.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
peri-implant plaque | 3 years
  modified plaque index
peri-implant bleeding | 3years
  bleeding index
peri-implant probing depth | 3 years
  measurements of probing depth in mm
overdenture retention | 3 years
  Measurements of retention values: using the device of measuring the clinical retentive forces
patient satisfaction | 3 years
  Assessment of patient satisfaction and Oral Health-Related Quality of Life: using a visual analog scale (VAS) questionnaire

SECONDARY OUTCOMES:
bone loss | 3 years
  evaluation of the peri-implant bone loss in mm

CONTACTS AND LOCATIONS:
Overall Officials: Khloud Ezzat, PhD, Principal Investigator — Lecturer
Locations (1):
- Khloud Ezzat, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No